CLINICAL TRIAL: NCT05069155
Title: Gamification to Improve Physical Activity in Older Adults at Risk for Alzheimer's: the STEP 4Life Trial
Brief Title: The STEP 4Life Trial
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Pennsylvania (Other)
Collaborators: National Institute on Aging (NIA) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Health Services Research
Other Study IDs: 849329; 5P30AG012836-20 (NIH)
Record Dates: First submitted 2021-07-08; First posted 2021-10-06 (Actual); Results first posted 2023-11-28 (Actual); Last update posted 2023-11-28 (Actual); Status verified 2023-11

CONDITIONS: Alzheimer Disease, At Risk; Alzheimer Disease, Protection Against; Dementia
Keywords: Alzheimers Disease; Gamification; Physical activity; Behavioral Science
MeSH Terms: conditions — Alzheimer Disease; Dementia; Motor Activity

STUDY DESIGN:
Intervention Model Description: This is a 2-arm, randomized, controlled trial over 12 weeks with 6 weeks of follow-up (18 weeks total) that compares a control group that uses a wearable device to track physical activity to an intervention group that uses the same wearable devices and receives a supportive social incentive-based gamification intervention to adhere to a step goal program.
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control (No Intervention): Participants will receive a wearable device (e.g. FitBit) but no other interventions during the intervention or follow-up periods.Participants will also complete milestones within the study, such as the cognition and function assessment during weeks 1- 2, and 15-16. Participants will complete an end-of-study questionnaire on their experience with the wearable device and time in the study.
- Gamification (Experimental): Intervention participants will receive a wearable device (e.g. FitBit) and will enter a game designed with behavioral economics concepts to address predictable barriers to behavior change during a 12-week intervention period.
  At the end of the 12 week intervention period, participants will enter a 6 week follow-up period during which interventions will cease but passive data collection of step counts will continue. Participants will also complete milestones within the study, such as the cognition and function assessment during weeks 1- 2, and 15-16. Participants will complete an end-of-study questionnaire on their experience with the wearable device and intervention design.
  Interventions: Behavioral: Gamification

INTERVENTIONS:
Behavioral: Gamification — Each participant signs a pre-commitment contract agreeing to try their best to achieve their daily step goal. Each week over the 12 week intervention period, participants are endowed 70 points (10/day). Participants are informed they will lose 10 points for each day the step goal is not met. Points are replenished at the start of the week. At the end of the week, if the participant has 40 points or more, he/she will advance one level, or drop one level if they have less than 40 points. The levels include: blue (lowest), bronze, silver, gold, platinum (highest). Each participant begins in the middle (silver). Each participant will also select a spouse, family member, or friend that they see often to serve as a supportive sponsor that receives a weekly email participants progress including points, game level, and average step countThis supportive sponsor will help to enhance social incentives to motivate the individual towards his or her goal.
  Arms: Gamification

SUMMARY:
The objective of this study is to test the feasibility of using behavioral economic interventions (gamification with social incentives) targeting daily step counts to prevent or delay the development of Alzheimer's Disease and Related Dementias (ADRD).

DETAILED DESCRIPTION:
Increased physical activity by walking further or more vigorously may prevent or delay the development of Alzheimer's Disease and Related Dementias (ADRD) but reaching higher levels of activity and maintaining it as a long-term habit is difficult to do. This project will use concepts from behavioral science to create a game older adults can play in order to increase their levels of activity while having fun doing it. The game is played with a support partner who is a spouse, family member, or close friend who provides feedback and encouragement to help the game-player reach activity goals and maintain them as habits over time. Participants in the game will use their own smartphone and a wristwatch that tracks activity (such as a FitBit, provided by this study) to set goals, get feedback, and play the game for 12 weeks. Participants will be asked to continue wearing the wristwatch for another 6 weeks to track activity after the game is over. To determine the effectiveness of this game, investigators will randomly assign 50 people to the game and 50 people to only get the wristwatch but no game component. All participants in this study will be recruited from an online registry of adults age 55-75 who have not been diagnosed with Alzheimer's (GeneMatch) which offers genetic testing on risk for ADRD to all participants. Investigators will recruit participants who have elevated genetic risk as well as those without specific genetic risks for the study to see if either group responds differently to the game.

ELIGIBILITY:
Inclusion Criteria:

* own a smartphone
* be enrolled in GeneMatch
* know their genetic testing results (APOE4)
* able to provide informed consent

Exclusion Criteria:

* Inability to provide informed consent
* does not have daily access to a smartphone compatible with the wearable device and not willing to use a device that we can provide them
* already enrolled in another physical activity study
* unable to ambulate independently
* any other medical conditions that would prohibit participation in physical activity program

Ages: 55 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 240 (Actual)
Dates: Start 2021-11-01 (Actual); Primary Completion 2022-11-21 (Actual); Study Completion 2023-01-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ryan Greysen, MD, MHS, MA, Principal Investigator — University of Pennsylvania
Locations (1):
- Blockley Hall, Philadelphia, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No
Individual participant data will not be made available.

REFERENCES:
- [Derived] Greysen SR, Oon AL, Harkins K, Rareshide C, Mondal A, Patel MS, Grill JD, Karlawish J. Effect of gamification with a support partner to increase physical activity in older adults at risk for Alzheimer's disease: The STEP 4Life randomized clinical trial. Alzheimers Dement. 2024 Aug;20(8):5450-5459. doi: 10.1002/alz.14058. Epub 2024 Jul 4. PMID 38962958

RESULTS

PARTICIPANT FLOW:
Recruitment Details: After a participant consented to participating in the study, they are given a Fitbit device to wear for a 2 week run-in period to collect step and sleep data to estimate their 2-week baseline. Participants with a baseline above 7500 are excluded from the study due to them being too active.
Pre-assignment Details: 240 participants were officially consented and enrolled per study design protocol. Out of 240, 137 are deemed ineligible due to high baseline (>7500 steps) during the 2-week run-in or did not complete all recruitment steps before the study closed for enrollment.
  Out of 103 randomized, 9 from the intervention arm dropped before starting the study.
Groups:
- Gamification: Intervention participants will receive a wearable device (eg. FitBit) and enter a game designed with behavioral economics concepts over a 12-week intervention period. At the end of the 12 weeks, participants will enter a 6 week follow-up period where interventions will cease but passive step data collection will continue. Participants will complete milestones within the study: cognition and function assessment at weeks 1- 2, and 15-16. They will complete an end-of-study questionnaire on their experience with the wearable device and intervention design.
  Gamification: Each participant signs a pre-commitment contract agreeing to try their best to achieve their daily step goal. Each week over the 12 week intervention period, participants are endowed 70 points (10/day). Participants are told they will lose 10 points for each day the step goal is not met. Points are refreshed at the start of the week. At the end of the week, if the participant has 40 points or more, they will advance one level, or drop one level if they have less than 40 points. The levels include: blue (lowest), bronze, silver, gold, platinum (highest). Each participant begins in the middle (silver). Each participant will select a spouse, family member, or friend they see often to serve as supportive sponsor that receives a weekly email on participant progress including points, game level, and average step count. The supportive sponsor will enhance social incentives to motivate the participant towards their goal.
Period: Overall Study
Arm/Group | Control | Gamification
Started | 50 | 44
Completed | 49 | 41
Not Completed | 1 | 3
Not completed — Withdrawal by Subject | 1 | 3

BASELINE CHARACTERISTICS:
Population: 94 participants were started in the study, but 4 participants dropped out. 90 participants completed the entire study.
Groups:
- Total: Total of all reporting groups
Arm/Group | Control | Gamification | Total
Number analyzed (Participants) | 50 | 44 | 94
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 1 | 2 | 3
  >=65 years | 49 | 42 | 91
Sex: Female, Male [Count of Participants; unit: Participants] — Population: Larger amount of participants in intervention arm dropped out or considered lost to follow-up compared to control arm.
  Participants
    Female | 36 | 34 | 70
    Male | 14 | 10 | 24
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants] — Population: Larger amount of participants in intervention arm dropped out or considered lost to follow-up compared to control arm.
  Participants
    Hispanic or Latino | 0 | 2 | 2
    Not Hispanic or Latino | 50 | 42 | 92
    Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants] — Population: Larger amount of participants in intervention arm dropped out or considered lost to follow-up compared to control arm.
  Participants
    American Indian or Alaska Native | 1 | 0 | 1
    Asian | 1 | 0 | 1
    Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
    Black or African American | 0 | 0 | 0
    White | 48 | 44 | 92
    More than one race | 0 | 0 | 0
    Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants] — Population: Larger amount of participants in intervention arm dropped out or considered lost to follow-up compared to control arm.
  Participants
    United States | 50 | 44 | 94
APOE4 genotype [Count of Participants; unit: Participants] — The APOE4 genotype increases the risk of developing Alzheimer's disease. Participants are categorized as being a carrier (higher risk) or non-carrier.
  Participants
    Carrier | 26 | 26 | 52
    Non-carrier | 23 | 17 | 40
    Missing | 1 | 1 | 2

OUTCOME MEASURES:

1. Primary Outcome: Change in Mean Daily Steps From the Baseline Period to the End of the 12 Week Intervention Period.
Description: The primary outcome of the study is the change in mean daily steps from the baseline period to the end of the 12 week intervention period collected by Fitbit Inspire device.
Time Frame: Baseline to 12 week intervention period (Weeks 1 - 12)
Measure: Mean (Standard Deviation); unit: steps
Arm/Group | Control | Gamification
Number analyzed (Participants) | 50 | 44
steps | 735 (1306) | 2422 (1460)

2. Secondary Outcome: Change in Mean Daily Step Counts During the 6 Week Follow-up Period After the End of the Intervention Period Tracked by Fitbit Inspire Device.
Description: The secondary outcome will examine the change in mean daily step counts during the 6 week follow-up period after the end of the 12 week intervention period.
Time Frame: 6 week follow-up period (Weeks 13 - 18)
Measure: Mean (Standard Deviation); unit: steps
Arm/Group | Control | Gamification
Number analyzed (Participants) | 50 | 44
steps | 705 (1916) | 1983 (1478)

3. Other Pre Specified Outcome: Change in Moderate-vigorous Physical Activity Minutes (MVPA) During the Start of the Intervention Period Compared to Baseline Period.
Description: MVPA is defined as ≥ 100 steps per minute. We will calculate minutes of MVPA per day.
Time Frame: Baseline to 12 week intervention period (Weeks 1-2)
Measure: Mean (Standard Deviation); unit: minutes
Arm/Group | Control | Gamification
Number analyzed (Participants) | 50 | 44
minutes | 4.2 (6.4) | 9.1 (10.4)

4. Other Pre Specified Outcome: Change in Moderate-vigorous Physical Activity (MVPA) Minutes During the Baseline and Follow-up Period (Weeks 13-18).
Description: MVPA is defined as ≥ 100 steps per minute. We will calculate minutes of MVPA per day.
Time Frame: Baseline and 6 week follow-up period (Weeks 13 - 18)
Measure: Mean (Standard Deviation); unit: minutes
Arm/Group | Control | Gamification
Number analyzed (Participants) | 50 | 44
minutes | 3.8 (11.5) | 8 (11.9)

ADVERSE EVENTS:
Time Frame: 12-week intervention and 6-week follow-up
Arm/Group | Control | Gamification
All-Cause Mortality (participants affected / at risk) | 0/50 | 0/44
Serious Adverse Events (participants affected / at risk) | 0/50 | 0/44
Other Adverse Events (participants affected / at risk) | 2/50 | 2/44
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Control (N=50) | Gamification (N=44)
Skin rash (Skin and subcutaneous tissue disorders) | 2 (2) | 2 (2) — Rash at the site of watch wristband

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-06-03): https://cdn.clinicaltrials.gov/large-docs/55/NCT05069155/Prot_SAP_000.pdf